CLINICAL TRIAL: NCT06358092
Title: Spleen Stiffness and Liver Stiffness Measured by Two-dimensional Shear Wave Elastography for Assessment of Cirrhosis and Portal Hypertension
Brief Title: Two-dimensional Shear Wave Elastography for Assessment of Cirrhosis and Portal Hypertension
Status: Not yet recruiting | Type: Observational
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yifei Huang, Doctor, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: ZSSYXHNK2401
Record Dates: First submitted 2024-03-29; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Cirrhosis, Liver; Portal Hypertension
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: To explore the cut-off value of LSM and SSM by 2D-SWE for assessment of CSPH in cirrhosis.
  Interventions: Diagnostic Test: Hepatic venous pressure gradient; Diagnostic Test: Two-Dimensional Shear Wave Elastography
- Validation cohort: To validate the cut-off value of LSM and SSM by 2D-SWE for assessment of CSPH in cirrhosis.
  Interventions: Diagnostic Test: Hepatic venous pressure gradient; Diagnostic Test: Two-Dimensional Shear Wave Elastography

INTERVENTIONS:
Diagnostic Test: Hepatic venous pressure gradient — HVPG is a measurement used to assess portal hypertension, a condition characterized by increased blood pressure in the portal vein, which carries blood from the digestive organs to the liver. HVPG measurement involves inserting a catheter into the hepatic vein via jugular vein puncture to directly measure the pressure within the liver. By comparing the pressure in the hepatic vein with that in the portal vein, HVPG provides valuable information about the severity of portal hypertension and helps in predicting clinical outcomes in patients with liver cirrhosis and related conditions. HVPG measurements are crucial in guiding treatment decisions, assessing treatment response, and predicting the risk of complications such as variceal bleeding and liver failure.
Diagnostic Test: Two-Dimensional Shear Wave Elastography — 2D-SWE is a non-invasive imaging technique used to assess tissue stiffness, particularly in the liver. This technology utilizes ultrasound to generate shear waves within the tissue being examined. By measuring the speed of these shear waves as they propagate through the tissue, 2D-SWE can provide quantitative information about tissue elasticity or stiffness. In the context of liver disease, including cirrhosis and fibrosis, 2D-SWE is valuable for evaluating the degree of liver stiffness, which correlates with the severity of liver fibrosis. This information aids in diagnosis, staging, and monitoring of liver diseases, allowing for early detection of complications and assessment of treatment response. Compared to traditional biopsy-based methods, 2D-SWE offers the advantage of being non-invasive, rapid, and repeatable, making it a preferred modality for assessing liver stiffness in clinical practice.

SUMMARY:
Exploring and establishing new non-invasive risk stratification techniques for portal hypertension based on E imaging technology for measuring liver and spleen stiffness is an urgent need in this field of research.

DETAILED DESCRIPTION:
Portal hypertension is an important risk factor affecting the clinical prognosis of patients with liver cirrhosis. According to clinical practice guidelines, risk stratification based on portal vein pressure levels is crucial for predicting the prognosis of patients with cirrhotic portal hypertension, and it is one of the most important aspects in the diagnosis and treatment chain of end-stage liver diseases such as cirrhosis. The most reliable method for assessing portal vein pressure in patients with cirrhosis is the measurement of hepatic venous pressure gradient (HVPG). This is achieved by inserting a catheter into the hepatic vein via jugular vein puncture, measuring the free and wedged pressures, and calculating the difference to obtain HVPG. HVPG provides important information regarding treatment response, complication risks, and long-term prognosis for patients with cirrhotic portal hypertension: HVPG ≥ 10mmHg indicates an increased risk of varices, decompensation events, and hepatocellular carcinoma in compensated cirrhosis patients, HVPG ≥ 12mmHg is a high-risk factor for variceal bleeding, HVPG ≥ 16mmHg suggests an increased risk of death in patients with cirrhotic portal hypertension, and HVPG ≥ 20mmHg indicates higher failure rates of hemostatic treatment and increased mortality risk in patients with acute variceal bleeding. However, there are some issues with measuring HVPG, including invasiveness, technical requirements, and high costs, which limit its clinical application. The development of non-invasive assessment techniques for portal hypertension in cirrhosis has always been a hotspot and difficulty in this field.

In recent years, with the rapid development of ultrasound elastography technology, it has also been widely used in the field of liver diseases. Transient elastography, point shear wave elastography, and two-dimensional shear wave elastography (referred to as E imaging) all have important value in the non-invasive assessment of portal hypertension in cirrhosis. Ultrasound elastography, due to its advantages of non-invasiveness, rapidity, ease of operation, repeatability, safety, and ease of follow-up monitoring, is of great significance in risk stratification, precise management, and efficacy evaluation of portal hypertension in cirrhosis. Although liver stiffness has been applied in the diagnosis, treatment, and prognosis assessment of cirrhotic portal hypertension, transient elastography is still the main ultrasound elastography technique used clinically, and there are relatively few original studies related to spleen stiffness. Therefore, there is currently a lack of high-level clinical evidence based on E imaging technology for evaluating portal hypertension in cirrhosis in China, as well as a lack of original research on spleen stiffness assessment in cirrhotic portal hypertension.

In summary, exploring and establishing new non-invasive risk stratification techniques for portal hypertension based on E imaging technology for measuring liver and spleen stiffness is an urgent need in this field of research.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old;
2. Clinical diagnosis of liver cirrhosis (confirmed by pathological biopsy, imaging findings, or occurrence of relevant complications);
3. Scheduled for hepatic venous pressure gradient (HVPG) examination;
4. Planned to undergo measurement of liver and spleen stiffness using E imaging technology;
5. Voluntary signing of informed consent form.

Exclusion Criteria:

1. Contraindications to hepatic venous pressure gradient examination;
2. Liver intervention surgery scheduled between E imaging examination and HVPG examination;
3. Interval between E imaging examination and HVPG examination exceeds 14 days;
4. Presence of liver cancer;
5. Concurrent active, severe, life-threatening diseases;
6. History of the following surgeries: ① Transjugular intrahepatic portosystemic shunt (TIPS) procedure; ② Hepatectomy; ③ Splenectomy; ④ Liver transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis and portal hypertension
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
the diagnostic performance of liver and spleen stiffness by E imaging technology for clinically significant portal hypertension | 1 year
  Using HVPG as the gold standard, the diagnostic performance of measuring liver and spleen stiffness based on E imaging technology for clinically significant portal hypertension.

SECONDARY OUTCOMES:
the diagnostic performance of microvessel imaging of hepatic microcirculation by E imaging technology for clinically significant portal hypertension | 1 year
  Using HVPG as the gold standard, the diagnostic performance of microvessel imaging of hepatic microcirculation based on E imaging technology for clinically significant portal hypertension.
the difference among left, middle and right hepatic venous pressure gradient | 1 year
  the difference among left, middle and right hepatic venous pressure gradient

CONTACTS AND LOCATIONS:
Overall Officials: Bin Wu, Professor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Franchis R, Bosch J, Garcia-Tsao G, Reiberger T, Ripoll C; Baveno VII Faculty. Baveno VII - Renewing consensus in portal hypertension. J Hepatol. 2022 Apr;76(4):959-974. doi: 10.1016/j.jhep.2021.12.022. Epub 2021 Dec 30. PMID 35120736
- [Result] Kaplan DE, Ripoll C, Thiele M, Fortune BE, Simonetto DA, Garcia-Tsao G, Bosch J. AASLD Practice Guidance on risk stratification and management of portal hypertension and varices in cirrhosis. Hepatology. 2024 May 1;79(5):1180-1211. doi: 10.1097/HEP.0000000000000647. Epub 2023 Oct 23. No abstract available. PMID 37870298
- [Result] Dajti E, Ravaioli F, Zykus R, Rautou PE, Elkrief L, Grgurevic I, Stefanescu H, Hirooka M, Fraquelli M, Rosselli M, Chang PEJ, Piscaglia F, Reiberger T, Llop E, Mueller S, Marasco G, Berzigotti A, Colli A, Festi D, Colecchia A; Spleen Stiffness-IPD-MA Study Group. Accuracy of spleen stiffness measurement for the diagnosis of clinically significant portal hypertension in patients with compensated advanced chronic liver disease: a systematic review and individual patient data meta-analysis. Lancet Gastroenterol Hepatol. 2023 Sep;8(9):816-828. doi: 10.1016/S2468-1253(23)00150-4. Epub 2023 Jul 18. PMID 37478880